CLINICAL TRIAL: NCT01002898
Title: Treatment Outcomes and Plasma Level of Ritonavir-boosted Lopinavir Monotherapy Among HIV-infected Patients Who Had Non-nucleoside Reverse Transcriptase Inhibitor (NRTI) and NNRTI Failure: A Pilot Study
Brief Title: Ritonavir-boosted Lopinavir Monotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bamrasnaradura Infectious Diseases Institute (Other Government)
Responsible Party: Bamrasnaradura Infectious Diseases Institute, Bamrasnaradura Infectious Diseases Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4/2551
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2009-10

CONDITIONS: HIV
Keywords: HIV-1 RNA; Treatment experienced
MeSH Terms: interventions — Lopinavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lopinavir/ritonavir (Experimental)
  Interventions: Drug: lopinavir/ritonavir soft gel capsule

INTERVENTIONS:
Drug: lopinavir/ritonavir soft gel capsule — Ritonavir-boosted lopinavir in soft gel formulation at 400/100 mg and lamivudine at 150 mg were given twice daily.
  Other Names: Kaletra

SUMMARY:
To assess 48-week treatment responses, tolerability, and steady-state minimum plasma concentrations of ritonavir-boosted lopinavir monotherapy for salvage therapy in HIV-1 infected patients who failed antiretroviral regimens containing NRTI and NNRTI.

DETAILED DESCRIPTION:
Currently, non-nucleoside reverse transcriptase inhibitor (NNRTI)-based highly active antiretroviral therapy (HAART) is widely prescribed as an initial therapy for treatment naïve HIV-infected patients, particularly in many resource-constrained countries. However, in patients who have delayed detection of treatment failure in this setting, the virus is often resistant to most existing nucleoside reverse transcriptase inhibitors (NRTIs) and NNRTIs even failing from the first regimen. As a consequence, constructing the potent salvage regimens that combined 2 or 3 fully active drugs from existing drug classes is often impossible in many resource-constrained countries where new agents, such as integrase inhibitor and chemokine receptor antagonist, are neither available nor affordable. Nevertheless, the goal of attaining undetectable plasma HIV-1 RNA is remain mandatory. To date, several clinical studies derived from the western countries that included 2 or more active drugs clearly demonstrate effective therapeutic strategies for antiretroviral (ARV)-experienced HIV-1 infected patients. Hence, using ritonavir-boosted protease inhibitor in a salvage therapy was considered to be an option in the resource-constrained countries and the limitations of remaining active NRTIs usually lead to ritonavir-boosted protease inhibitor monotherapy as a salvage regimen.

Among several previous reports using ritonavir-boosted protease inhibitor, ritonavir-boosted lopinavir monotherapy has been extensively studied so far. Different strategies of ritonavir-boosted lopinavir monotherapy have been explored; however, most related clinical trials studied this regimen as either a treatment simplification strategy or induction therapy in treatment-naïve patients. A strategy to use ritonavir-boosted lopinavir monotherapy as a salvage regimen is not available. On the other hand, previous studies showed that continuation of lamivudine after emerging of the M184V mutation had somewhat benefit on immunological response and clinical progression in patients who had limited options of salvage regimens. Moreover, there is neither additional any other mutation nor increase resistance to other antiretroviral drugs. Thus, this is the reason why we added lamivudine to decrease viral fitness in the study regimen. The objective of this study was to assess 48-week treatment responses, tolerability, and steady-state minimum plasma concentrations of ritonavir-boosted lopinavir monotherapy for salvage therapy in HIV-1 infected patients who failed antiretroviral regimens containing NRTI and NNRTI.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infected patients >18 years of age,
2. failed NNRTI-based antiretroviral therapy with M184V, thymidine analogue mutations (TAMs) and NNRTI-associated mutations
3. had plasma HIV-1 RNA >1,000 copies/mL.

Exclusion Criteria:

1. Had a history of exposure to protease inhibitor
2. Receipt a medication that has drug-drug interactions with lopinavir.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To assess 48-week treatment responses of ritonavir-boosted lopinavir (LPV/r) monotherapy as salvage regimen. | 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Bamrasnaradura Infectious Diseases Institute, Nonthaburi, Changwat Nonthaburi, Thailand